CLINICAL TRIAL: NCT06716203
Title: A Randomized, Double-blind, Placebo-Controlled Trial Comparing the Efficacy and Safety of BGM0504 Versus Placebo in Patients with Type 2 Diabetes, Inadequately Controlled with Diet and Exercise Alone
Brief Title: A Study of BGM0504 in Poorly Controlled Type 2 Diabetes Patients Only Through Diet and Exercise
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BrightGene Bio-Medical Technology Co., Ltd. (Industry)
Collaborators: BrightGene New Bio-Medical Technology(Wuxi) Co.Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BGM0504-Ⅲ -T2DM-01
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental: 5 mg BGM0504 (Experimental): Experimental: 5 mg BGM0504 5 milligrams (mg) BGM0504 administered subcutaneously (SC) once a week.
  Interventions: Drug: Drug: 5 mg BGM0504 Administered SC
- Experimental: 10 mg BGM0504 (Experimental): Experimental: 10 mg BGM0504 10 mg BGM0504 administered SC once a week.
  Interventions: Drug: Drug: : 10 mg BGM0504 Administered SC
- Placebo Comparator: Placebo (Placebo Comparator): Placebo Comparator: Placebo Placebo administered subcutaneously (SC) once a week.
  Interventions: Drug: Drug: Placebo Administered SC

INTERVENTIONS:
Drug: Drug: 5 mg BGM0504 Administered SC — Drug: BGM0504 Administered SC
  Arms: Experimental: 5 mg BGM0504
Drug: Drug: : 10 mg BGM0504 Administered SC — Drug: BGM0504 Administered SC
  Arms: Experimental: 10 mg BGM0504
Drug: Drug: Placebo Administered SC — Drug: Placebo Administered SC
  Arms: Placebo Comparator: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled phase III clinical study to evaluate the efficacy and safety of BGM0504 in patients with type 2 diabetes (T2D) with poor glycemic control only through diet and exercise.

The main purpose is to evaluate the clinical efficacy of BGM0504 injection monotherapy for 32 weeks compared with placebo in Chinese patients with type 2 diabetes with poor glycemic control only through diet and exercise, and to evaluate the clinical efficacy and safety of BGM0504 injection for 52 weeks of administration.

ELIGIBILITY:
Inclusion Criteria:

* ☑ Have been diagnosed with type 2 diabetes mellitus (T2DM);

  * Have a BMI ≥23 kilograms per meter squared (kg/m²) at screening;
  * Be of stable weight (± 5%) for at least 3 months before screening;
  * Have HbA1c between ≥7.5% and ≤11.0%；
  * Fasting Plasma Glucose (FPG) ≤ 15.0 mmoL/L.

Exclusion Criteria:

* ■ Previous diagnosis of type 1 diabetes, special type diabetes ;

  * There are malignant tumors within 5 years before screening, or patients are in latent of clinical malignant tumors (except patients with skin basal cell carcinoma and squamous cell carcinoma, cervical carcinoma in situ, prostate carcinoma in situ or papillary thyroid carcinoma who have no recurrence after surgery).
  * Have had chronic or acute pancreatitis any time prior to study entry;
  * Known allergic constitution (allergy to 3 or more kinds of food or drugs), or allergy to GLP-1 receptor agonists, or severe allergic diseases (asthma, urticaria, eczematous dermatitis, etc.) at screening;
  * Mentally incapacitated or speech-impaired;
  * Suspected or confirmed history of alcohol or drug abuse;
  * Pregnant or lactating woman;
  * The investigator considers that there are any other conditions that make it inappropriate to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-12-29 (Estimated); Study Completion 2026-08-25 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Hemoglobin A1c (HbA1c) | Week 0 to Week 32
  Change from baseline in HbA1c after 32 weeks of treatment.

SECONDARY OUTCOMES:
Change From Baseline in Body Weight | Week 0 to Week 52
  Change from baseline in body weight after 52 weeks of treatment.
Change From Baseline in Hemoglobin A1c (HbA1c) | Week 0 to Week 52
  Change from baseline in HbA1c after 52weeks of treatment.
Percentage of Participants With HbA1c Target Value of <7% | Week 0 to Week 52
  Percentage of Participants With HbA1c Target Value of <7% after 52weeks of treatment.
Percentage of Participants With HbA1c Target Value of <5.7% | Week 0 to Week 52
  Percentage of Participants With HbA1c Target Value of <5.7%after 52weeks of treatment.
Change From Baseline in Fasting Serum Glucose | Week 0 to Week 52
  Change from baseline in FPG after 52 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China